CLINICAL TRIAL: NCT01308658
Title: A Phase I, Open-label, Randomized, 2-panel, 2-way Crossover Pivotal Bioequivalence Trial Between the Commercially Available 400-mg Tablet Formulation (F030) and the 800-mg Tablet Formulation of Darunavir (G002), in the Presence of Low-dose Ritonavir Under Fasted and Fed Conditions
Brief Title: TMC114-TiDP3-C176 - A Study in Healthy Volunteers Investigating the Bioequivalence Between Two Commercially Available 400-mg Tablets to One New 800-mg Tablet of Darunavir (DRV) in the Presence of Low-dose Ritonavir Under Fed and Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017776; TMC114-TiDP3-C176
Record Dates: First submitted 2011-02-03; First posted 2011-03-04 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: TMC114-C176; TMC114; DRV; HIV; Healthy volunteers
MeSH Terms: interventions — Darunavir; Ritonavir

ARMS (2):
- 001 (Experimental): Darunavir (DRV) 2x400-mg DRV tablet or 800-mg tablet on Day 3
  Interventions: Drug: Darunavir (DRV)
- 002 (Experimental): ritonavir 100-mg once daily on Day 1 to Day 5
  Interventions: Drug: ritonavir

INTERVENTIONS:
Drug: Darunavir (DRV) — 2x400-mg DRV tablet or 800-mg tablet
  Arms: 001
Drug: ritonavir — on Day 3
  Arms: 002

SUMMARY:
In this study participants will be given 800 mg darunavir, either as one 800-mg tablet formulation (G002), or as two commercially available 400-mg tablets formulation (F030), to evaluate the effect between both, in the presence of low-dose ritonavir under fasted and fed conditions.

DETAILED DESCRIPTION:
Darunavir (DRV, formerly known as TMC114) is an inhibitor of human immunodeficiency virus (HIV) protease. This study is designed to establish the bioequivalence of a commercially available 400-mg tablet formulation (F030) to one 800-mg tablet formulation of DRV (G002) in the presence of low-dose ritonavir under fasted and fed conditions. This is a Phase I, open-label (both participant and investigator know the name of the medication given at certain moment), randomized (study medication is assigned by chance), 2-panel, 2-way crossover study in healthy volunteers to assess the bioequivalence of DRV following administration of 2 tablet strengths (in the presence of low-dose ritonavir) under fasted and fed conditions. A total of 124 participants will participate in this study. Participants will be divided into 2 panels; 80 participants in Panel 1 (fasted) and 44 in Panel 2 (fed). In Panel 1, during 2 subsequent sessions, each participant will receive 2 treatments under fasted conditions, meaning Treatment A, a single oral 800-mg dose of DRV formulated as the 400-mg commercially available tablet F030 and Treatment B, a single oral 800-mg dose of DRV formulated as the 800-mg tablet formulation G002. In Panel 2, the same design as Panel 1 will be followed but under fed conditions, and where the 2 treatments, respectively, will be called Treatments C and D. In both panels, participants will receive ritonavir 100 mg once a day on Days 1 to 5. Ritonavir will be administered under fed conditions in both panels except for the morning intake on Day 3 in Panel 2 where it will be administered under fasting conditions. A washout period of at least 7 days between subsequent treatments will be observed. Safety (blood and urine tests, blood pressure, pulse, electrocardiogram, and physical examination) and tolerability evaluations will be recorded at regular intervals throughout the trial. Panel 1 (fasted condition) and Panel 2 (fed condition): a single dose of 800 mg DRV on Day 3 and 100 mg ritonavir once daily from Day 1 to 5. DRV will be formulated as the commercially available 400-mg tablet formulation (F030) or as the investigational 800-mg tablet formulation (G002). Ritonavir will be used as the commercially available melt-extrusion tablet containing ritonavir eq. 100 mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy based on a medical evaluation including medical history, physical examination, blood tests and electrocardiogram
* Body Mass Index of 18.0 to 30.0 kg/m² and non-smoker or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months
* Women must be postmenopausal for at least 2 years or be surgically sterile or be not heterosexually active for the duration of the study or have a vasectomized partner
* Men must agree to use a highly effective method of birth control.

Exclusion Criteria:

* Infection with Hepatitis A, B, or C virus
* infection with HIV
* Women who are pregnant or breastfeeding
* History of, or any current medical condition which could impact the safety of the participant in the study
* Previously participated in a multiple-dose study with DRV.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2011-01; Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of 100-mg ritonavir after a multiple oral dose on Days 1 to 5 in healthy volunteers in fed or fasted conditions | measured on Day 1 to Day 6
Plasma concentrations of Darunavir (DRV) after a single oral dose of 800-mg DRV on Day 3 in healthy volunteers in fed or fasted conditions | measured on Day 1
Plasma concentrations of DRV after a single oral dose of 800-mg DRV on Day 3 in healthy volunteers in fed or fasted conditions | measured on Day 3 to Day 6

SECONDARY OUTCOMES:
Incidence of all adverse events by treatment group | Measured from Day 1 until end of trial
Blood tests | Measured from Day 1 until end of trial
Measurements of blood pressure | Measured from Day 1 until end of trial
Measurements of pulse | Measured from Day 1 until end of trial
Measurements of electrocardiograms | Measured from Day 1 until end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (1):
- Berlin, Germany

REFERENCES:
- [Derived] Kakuda TN, Leopold L, Timmers M, Van De Casteele T, Hillewaert V, Tomaka FL, Hoetelmans RM. Bioavailability and bioequivalence of a darunavir 800-mg tablet formulation compared with the 400-mg tablet formulation. Int J Clin Pharmacol Ther. 2014 Sep;52(9):805-16. doi: 10.5414/cp202066. PMID 25109510